CLINICAL TRIAL: NCT00024492
Title: Study of Liposome Encapsulated Mitoxantrone (LEM) in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: INSYS Therapeutics Inc (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LEM-001
Record Dates: First submitted 2001-09-17; First posted 2001-09-18 (Estimated); Last update posted 2011-06-06 (Estimated); Status verified 2004-08

CONDITIONS: Tumors
Keywords: Liposome Encapsulated Mitoxantrone (LEM); solid tumors
MeSH Terms: conditions — Neoplasms

INTERVENTIONS:
Drug: Liposome Encapsulated Mitoxantrone (LEM)

SUMMARY:
Liposome entrapped mitoxantrone (LEM) is a mixture of commercially available mitoxantrone HCL (Novantrone) and a combination of lyophilized lipids. Mitoxantrone, the active agent in the investigational formulation, is a currently marketed chemotherapeutic agent. The rationale for development of liposomal formulations is primarily that of improving the safety profile of the drug, which may permit dose intensification and/or an increase in the cumulative dose that may be administered, resulting in enhanced efficacy.

LEM will be given to patients with advanced solid tumors to determine the dose of drug these patients can tolerate. Patients will receive intravenous LEM every 21 days until the disease progresses or toxicity occurs requiring treatment discontinuation. Anti-tumor effects of LEM will be assessed and patients will be evaluated for safety and tolerability.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose (MTD) and dose limiting toxicity (DLT) of LEM.

II. Measure the blood pharmacokinetics of LEM following IV administration.

III. Observe any anti-tumor effects of LEM.

PROTOCOL OUTLINE: This is an open-label study for patients with advanced and/or metastatic, histologically-documented solid tumors considered to be unresponsive to available conventional treatment.

LEM will be administered IV over 45 minutes. At least three patients will be studied at each dose level and at least three patients will complete one 21-day course before any patient is enrolled at the next dose level. Study drug administration will continue on an every 3-week schedule in the absence of progressive disease or unacceptable toxicity. A subsequent course of treatment may be administered at least 21 days after a prior LEM dose has been administered when study criteria are met.

Cohorts of 3 patients per dose level will be studied. This will be expanded to 6 if a DLT occurs, followed by a total of 6 patients at a possible MTD.

PROJECTED ACCRUAL: It is expected that 21 to 30 patients will be entered into the study to determine the MTD: 3 per dose level, expanded to 6 if DLT occurs, followed by a total of 6 patients at a possible MTD. The dose level identified as the MTD may then be expanded up to 12 patients to permit additional safety assessment.

ELIGIBILITY:
-Disease Characteristics-

Advanced (local and/or metastatic) histologically documented solid tumors

Disease is not considered responsive to available conventional modalities or treatments

-Prior/Concurrent Therapy-

Must be fully recovered from acute toxicities of any prior treatment with cytotoxic drugs, radiotherapy or other anti-cancer modalities (returned to baseline before most recent treatment)

No radiotherapy, treatment with cytotoxic or biologic agents within 3 weeks prior to study entry (6 weeks for mitomycin or nitrosoureas)

At least 2 weeks after any prior surgery or hormonal therapy

Chronic toxicities of grade 1 from prior treatment are permitted

-Patient Characteristics-

ECOG Performance status of 0-2

Must be at least 18 years of age

Must have the following clinical laboratory values: ANC at least 1,500/mm3; Platelets at least 100,000/mm3; Hemoglobin at least 10 g/dL; albumin at least 3.0 mg/dL; Serum creatinine at least 2.0 mg/dL; Total bilirubin not more than upper limit of normal; ALT, AST, and alkaline phosphatase not more than 1.5 x upper limit of normal; LVEF by MUGA scan greater than or equal to the lower limit of normal

Must sign informed consent

No pregnant and/or nursing patients. Women of child-bearing potential must have negative serum or urine pregnancy test within 1 week prior to study entry. Sexually-active patients (both men and women) must use acceptable contraceptive methods.

No active uncontrolled bleeding or bleeding diathesis (e.g., active peptic ulcer disease)

No active infection of any kind

No known HIV infection or viral hepatitis

No active heart disease including myocardial infarction within the previous 6 months, symptomatic coronary artery disease, arrhythmias requiring medication, or congestive heart failure

No known CNS metastases

No patients receiving any other standard or investigational treatment for their cancer, or any other investigational agent for any indication

No patients requiring immediate palliative treatment of any kind including surgery

No patients who have received a high-dose chemotherapy regimen with stem cell support in the previous 6 months

No patients who have received a cumulative anthracycline dose greater than 250 mg/m2 (doxorubicin equivalent)

No patients unwilling or unable to follow protocol requirements

No patients with known hypersensitivity to mitoxantrone or liposomes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2001-08; Study Completion 2004-06

CONTACTS AND LOCATIONS:
Overall Officials: Przemyslaw Twardowski, M.D., Principal Investigator — City of Hope National Medical Center
Locations (4):
- United States (4):
  - City of Hope National Medical Center, Duarte, California
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - The Ohio State University, Columbus, Ohio